CLINICAL TRIAL: NCT06723405
Title: A Randomized, Double-blind, Placebo-controlled, Proof-of-concept Study of EVO301 in Adults With Atopic Dermatitis
Brief Title: Efficacy Study of EVO301 in Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evommune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EVO301-AD001
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (AD); Eczema; Eczema Atopic Dermatitis
Keywords: atopic dermatitis; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous EVO301 (Experimental)
  Interventions: Biological: EVO301
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: EVO301 — Intravenous EVO301
  Arms: Intravenous EVO301
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2a efficacy and safety study of EVO301 for the treatment of adults with atopic dermatitis.

DETAILED DESCRIPTION:
This is a Phase 2a efficacy and safety study of intravenous EVO301 in adults with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-lactating females, age 18 years or older
2. Chronic atopic dermatitis for at least 6 months
3. BSA of AD involvement of at least 10%
4. EASI score of at least 16.

Exclusion Criteria:

1. Significant AD flare with 4 weeks
2. Use of biologic therapy within 12 weeks
3. Regular use of tanning booth within 4 weeks
4. Skin condition that could interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | 12 weeks
  EASI assesses the extent and severity of atopic dermatitis. EASI is a composite index with scores ranging from 0 to 72. Higher values indicate more severe or extensive disease.

SECONDARY OUTCOMES:
Investigator Global Assessment (IGA) | 12 weeks
  The IGA assesses the overall appearance and severity of atopic dermatitis using a 5-point scale [0 (clear) to 4 (severe)].
Body Surface Area (BSA) | 12 weeks
  BSA estimates the extent of atopic dermatitis involvement and is expressed as a percentage of total body surface area.
Pruritus-NRS | 12 weeks
  The pruritus-NRS is an 11-point scale used by subjects to rate their worst itch severity over the past 24 hours with 0 indicating "no itch" and 10 indicating "worst itch imaginable".

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (2):
  - Cornerstone Dermatology, Coorparoo
  - Momentum Clinical Research Darlinghurst, Darlinghurst
- New Zealand (10):
  - Pacific Clinical Research Network (PCRN) Auckland, Auckland
  - Optimal Clinical Trials North, Auckland
  - Optimal Clinical Trials, Auckland
  - Pacific Clinical Research Network (PCRN) Christchurch, Christchurch
  - Momentum Clinical Research Dunedin, Dunedin
  - Clinical Trials New Zealand Ltd, Hamilton
  - Momentum Clinical Research Lower Hutt, Hutt Central
  - Pacific Clinical Research Network (PCRN) Tasman, Nelson
  - Momentum Clinical Research Kapiti, Paraparaumu
  - Momentum Clinical Research Pukekohe, Pukekohe